CLINICAL TRIAL: NCT04969692
Title: Local Warming Technique for Arterial Cannulation in Adult Patients Under Heart Surgery-A Randomized Controlled Trial
Brief Title: Local Warming Technique for Arterial Cannulation in Adult Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Clinical associate professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 05-2021-117
Record Dates: First submitted 2021-07-08; First posted 2021-07-21 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Cardiac Disease Which Should be Treated by Surgery
MeSH Terms: interventions — Temperature

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-warming group (No Intervention): non-warming of local skin (puncture site)
- warming group (Active Comparator): warming to increase local skin (puncture site) temperature
  Interventions: Procedure: warming to increase local skin (puncture site) temperature

INTERVENTIONS:
Procedure: warming to increase local skin (puncture site) temperature — According to the group of participants, investigator applies the warmer to the hands and wrists of the participants, makes a local temperature of 40℃ gradually, and maintains it for about 10 minutes in warming group (which is divided in to warming-palpation (WP) and warming-US (WU) group).
  Arms: warming group

SUMMARY:
Based on the fact that arterial vasodilation can be advantageous for endovascular catheterization and that an increase in body temperature can cause vasodilation by activating the cholinergic active vasodilator system, this study was planned to observe whether there was a significant change in the diameter of artery through ultrasound and to confirm the effectiveness of heating in the traditional palpation technique and the US-guided technique after local warming of the insertion site of arterial catheter in adult patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
Arterial cannulation is one of the important clinical techniques commonly used for real-time monitoring of blood pressure changes or when repeated blood tests are required. However, complications such as bleeding, hematoma, and vascular occlusion may occur if the operator has little or no experience in the procedure, or if arterial cannulation is not easy due to the patient's underlying disease and systemic factors. This situation prolongs the anesthesia induction time and may cause great harm to the patient in cases with a high bleeding tendency, such as in cardiac surgery. Various studies have reported various arterial cannulation techniques so far, and there have been many advances in arterial cannulation techniques due to the general use of ultrasound (hereafter US). However, there is still a risk of complications due to inexperience in the use of US or poor vascular status of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age undergoing cardiac surgery under general anesthesia

Exclusion Criteria:

* If the patient already has an arterial catheter and does not need additional arterial cannulation.
* When arterial cannulation is performed on an artery other than the radial artery due to the surgical technique or the patient's condition.
* When the patient's condition is urgent, such as emergency surgery, and there is no time to proceed with the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-03-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
changes of the diameter of the artery | from time point of warming to success of arterial cannulation (the day of surgery, up to 1hour)
  Investigator measures where there is a significant increase in the diameter of the artery due to warming using US.
changes of the cross-sectional area of the artery | from time point of warming to success of arterial cannulation (the day of surgery, up to 1hour)
  Investigator measures where there is a significant increase in the cross-sectional area of the artery due to warming using US.
Success rate of first trial for arterial cannulation | from time point of warming to success of arterial cannulation (the day of surgery, up to 1hour)
  Investigator measures success rate of first trial for arterial cannulation.

SECONDARY OUTCOMES:
Complications related with arterial cannulation | from time point of warming to success of arterial cannulation (the day of surgery, up to 1hour)
  Investigator measures where there are complications such as hematoma, vasopasm, and ischemia.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, MD, PhD, Principal Investigator — Department of Anesthesia and Pain Medicine, School of Medicine, Pusan National University
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park S, Kim HJ, Heo W, Shin SW, Yoon JU, Byeon GJ, Lee J, Jung J, Kim HY. Effect of local warming for arterial catheterization in adult cardiac surgery: a randomized controlled trial. J Thorac Dis. 2023 Oct 31;15(10):5330-5339. doi: 10.21037/jtd-23-820. Epub 2023 Sep 18. PMID 37969298